CLINICAL TRIAL: NCT02858804
Title: EDOCH Alternating With DHAP Regimen Combined Rituximab or Not to Treat New Diagnosed Younger (Age≤65 Years) Mantle Cell Lymphoma in China: A Multicentre Phase III Trial
Brief Title: EDOCH Alternating With DHAP for New Diagnosed Younger MCL
Acronym: BDH-MCL01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015007
Record Dates: First submitted 2016-07-17; First posted 2016-08-08 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: mantle cell lymphoma; EDOCH; DHAP; maintenance therapy
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Etoposide; Doxorubicin; Dexamethasone; Vincristine; Cyclophosphamide; Cytarabine; Cisplatin; Rituximab; Thalidomide; Prednisone; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Etoposide (Experimental): 50 mg/m2, IV, d1-4
  Interventions: Drug: Etoposide
- Doxorubicin (Experimental): 10 mg/m2, IV, d1-4
  Interventions: Drug: Doxorubicin
- Dexamethasone (Experimental): 30 mg/d, d1-5
  Interventions: Drug: Dexamethasone
- Vincristine (Experimental): 0.4 mg/m2, IV, d1-4
  Interventions: Drug: Vincristine
- Cyclophosphamide (Experimental): 750 mg/m2 ,d5
  Interventions: Drug: Cyclophosphamide
- Cytarabine (Experimental): 2g/m2, q12h, d1
  Interventions: Drug: Cytarabine
- Cisplatin (Experimental): 100mg/ m2,IV, d1
  Interventions: Drug: Cisplatin
- Rituximab (Experimental): 375 mg/m2 IV, d1
  Interventions: Drug: Rituximab
- Thalidomide (Experimental): 50-150mg/d, po, d1-28
  Interventions: Drug: Thalidomide
- Prednisone (Experimental): 0.5mg/Kg, po, qod
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Etoposide — 50 mg/m2, IV d1-4
  Other Names: VP-16
  Arms: Etoposide
Drug: Doxorubicin — 10 mg/m2, IV, d1-4
  Other Names: adriamycin
  Arms: Doxorubicin
Drug: Dexamethasone — 30 mg/d, d1-5
  Other Names: Dex
  Arms: Dexamethasone
Drug: Vincristine — 0.4 mg/m2, IV, d1-4
  Other Names: VCR
  Arms: Vincristine
Drug: Cyclophosphamide — 750 mg/m2 ,d5
  Other Names: CTX
  Arms: Cyclophosphamide
Drug: Cytarabine — 2g/m2, q12h, d1
  Other Names: Ara-c
  Arms: Cytarabine
Drug: Cisplatin — 100mg/ m2,IV, d1
  Other Names: DDP
  Arms: Cisplatin
Drug: Rituximab — 375 mg/m2 IV, d1
  Other Names: R
  Arms: Rituximab
Drug: Thalidomide — 50-150mg/d, po, d1-28
  Other Names: Thal
  Arms: Thalidomide
Drug: Prednisone — 0.5mg/Kg, po, qod
  Other Names: Pred
  Arms: Prednisone

SUMMARY:
The purpose of this study is to:

1. determine the efficiency of EDOCH (etoposide,dexamethasone,doxorubicin, cyclophosphamide and vincristine) alternating with DHAP (cisplatin, cytarabine and dexamethasone) regimen combined with rituximab or not in young mantle cell lymphoma patients (age≤65 years);
2. determine the efficiency of rituximab and thalidomide plus prednisone as maintenance regimens.

DETAILED DESCRIPTION:
Enrolled patients will receive EDOCH (etoposide,dexamethasone,doxorubicin, cyclophosphamide and vincristine) ±R /DHAP(cisplatin, cytarabine and dexamethasone) ±R alternating chemotherapy. If a partial remission or better response achieves, patients will be recommended to receive autologous stem cell transplantation as consideration therapy or another two cycles EDOCH ±R /DHAP±R chemotherapy (based on patient's choice). Patients with less than partial remission (PR) response will quit this study. After treatments finished, maintenance therapy with rituximab or thalidomide plus prednisone will be given less than two years. The determination of maintenance regimens is dependent on patients choices.

ELIGIBILITY:
Inclusion Criteria:

* age≤65 years
* diagnosis with mantle cell lymphoma
* Ann Arbor stage II,III or IV
* ECOG≤1 or if ECOG≥2 but recover after pretreatment.

Exclusion Criteria:

* with centre neural system involvement
* serious complications such as uncontrolled diabetes, gastric ulcer or other serious angiocardiopathy determined by the physician
* HIV positive or active HBV infection or other uncontrolled systematic infection
* clinical central nervous dysfunction
* serious surgery within 30 days
* pregnancy or baby nursing period or un-contracepted child bearing period woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
progression free survival | up to 36 months
  the time interval between diagnosis and disease progression or death or last follow-up

SECONDARY OUTCOMES:
complete remission | up to 6 months
  measure with normal serum immunofixation electrophoresis and normal bone marrow feature, and without symptoms and enlarged organs
overall survival | up to 36 months
  time interval between diagnosis and death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Doc, Principal Investigator — Blood disease hospital, Chinese Academic Medical School
Locations (1):
- Shuhua Yi, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided